CLINICAL TRIAL: NCT04518787
Title: Genetic Biomarkers Associated With Child Language Development in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 201901976A3
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Child Language
Keywords: language development; gene; whole-exome sequencing; body function and body structure; quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Healthy child
- Experimental: Patients with language disorder

SUMMARY:
A study of the relation between genetic biomarkers and child language development in Taiwan.

DETAILED DESCRIPTION:
The interaction between gene and environment (G×E) can be a very complicated process that influences child development. As a pilot study of child development biomarkers, this study investigates genes related to child language development and language disorder.

ELIGIBILITY:
Inclusion Criteria of Healthy Child:

* Age 2-18 y/o
* Agree to sign informed consent

Exclusion Criteria of Healthy Child:

* Central nervous system disease
* Neuromuscular Disorders
* Congenital Abnormality
* Genetic Disease
* Dysesthesia
* Hearing Impairment

Inclusion Criteria of Child with language disorder:

* Patients with Language Disorder
* Age 2-18 y/o
* Agree to sign informed consent

Exclusion Criteria of Child with language disorder:

* Hearing Impairment

Inclusion Criteria of Adult:

* His or her child participated in this study, and gene abnormality was found.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Control and experimental groups
Sampling Method: Non-Probability Sample
Enrollment: 596 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Scores of cognitive function 1 | baseline
  Bayley Scales of Infant and Toddler Development (Scores from 0 to 140, higher scores mean a better outcome.)
Scores of cognitive function (2 y/o to 6 y/o) | baseline
  Wechsler Preschool and Primary Scale of Intelligence (Scores from 0 to 200, higher scores mean a better outcome.)
Scores of cognitive function (6 y/o to 16 y/o) | baseline
  Wechsler Intelligence Scale for Children (Scores from 0 to 200, higher scores mean a better outcome.)
Scores of cognitive function 3 | baseline
  Test of Nonverbal Intelligence-Fourth Edition (Scores from 0 to 60, higher scores mean a better outcome.)
Scores of language function 1 | baseline
  Peabody Picture Vocabulary Test-Revised (Scores from 0 to 124, higher scores mean a better outcome.)
Scores of language function 2 | baseline
  Preschool Language Impaired Scale(PLS)/Language Impaired Scale(LS) (PLS: Scores from 0 to 65, higher scores mean a better outcome. LS: Scores from 0 to 73, higher scores mean a better outcome.)
Scores of general development | baseline
  Comprehensive Developmental Inventory for Infants and Toddlers (Higher scores mean a better outcome.)
Gene test 1 | baseline
  Microarray (Use Axiom Genome-Wide TWB 2.0 Array Plate (TWB 2.0) to analyze SNPs of disease-related biomarkers.)
Gene test 2 | baseline
  Whole-Exome Sequencing (Use Burrows-Wheeler Aligner (BWA) 85, Samtools86, Picard, Genome Analysis Toolkit (GATK) to screen out the variant discovery and genotyping.)

SECONDARY OUTCOMES:
Scores of participation(2-5 y/o) | baseline
  Assessment of Preschool Children's Participation (Scores from 0 to 45, higher scores mean a better outcome.)
Scores of participation(>6 y/o) | baseline
  Children Assessment of Participation and Enjoyment and Preferences for Activity of Children (Higher scores mean a better outcome.)
Scores of activities | baseline
  Functional Independence Measure for Children (Scores from 18 to 126, higher scores mean a better outcome.)
Scores of quality of life | baseline
  Pediatric Quality of Life Inventory TM (Scores from 0 to 102, higher scores mean a better outcome.)

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, MD, PhD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No